CLINICAL TRIAL: NCT00587600
Title: Biomarkers in Phototherapy of Barrett's Esophagus
Acronym: BIOBAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kenneth K. Wang, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2138-00; CA97048-05
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Barrett's Esophagus; High Grade Dysplasia
Keywords: Barrett's Esophagus; High Grade Dysplasia; Photodynamic Therapy
MeSH Terms: conditions — Barrett Esophagus | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photodynamic therapy (Active Comparator): will have photodynamic therapy
  Interventions: Procedure: Photodynamic therapy
- radiofrequency ablation of barretts esophagus (Active Comparator): radiofrequency ablation of barretts esophagus
  Interventions: Procedure: radiofrequency ablation of barrett's esophagus

INTERVENTIONS:
Procedure: Photodynamic therapy — Photofrin 2mg/kg Photoradiation The light dose delivered will be a total of 200 joules per centimeter fiber which has previously been shown to ablate Barrett's mucosa.
  Arms: Photodynamic therapy
Procedure: radiofrequency ablation of barrett's esophagus — radiofrequency ablation
  Arms: radiofrequency ablation of barretts esophagus

SUMMARY:
This study is being done to find out if Photodynamic Therapy (treatment with a red light and a drug called photofrin) or Radiofrequency ablation works the same for patients who have biomarkers (abnormalities in molecules of cells that may or may not help predict cancer) present in their Barrett's esophagus as for patients who do not have biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have biopsy proven Barrett's esophagus with evidence of specialized intestinal epithelium and dysplasia (either high grade dysplasia or low grade dysplasia) on histology.
* Patients must have endoscopically visible segments of Barrett's esophagus of greater than 1 centimeter in length.
* All patients must be eligible for longterm follow-up as well as tolerate endoscopy, biopsy, and cytology.
* Patients must be willing to travel to Rochester, Minnesota for follow-up
* Patients must have a friend or relative accompany them on visits since sedatives will render them unable to operate a motor vehicle
* If patients are on anticoagulation, they must be able to tolerate reversal of anticoagulation for study biopsies and therapy
* All patients must be able to tolerate proton pump inhibitor therapy. Esomeprazole will be provided but can be changed to another proton pump inhibitor if the patient is intolerant.
* All patients who have histological or cytological evidence of high grade dysplasia will be seen by an experienced thoracic surgeon for consideration of esophagectomy.

Exclusion Criteria:

* Patients who are unable to follow light avoidance instructions
* Patients with a history of prior esophageal surgery or successful fundoplication
* Patients who had prior photodynamic therapy
* Patients with pre-existing strictures in their esophagus
* Patients who have known allergies to porphyrin compounds
* Patients with a prior biopsies of Barrett's esophagus that contain carcinoma
* Patients who require continuous anti-coagulation
* Patients who are pregnant or are capable of pregnancy will be excluded from this study unless they have been on effective birth control measures
* Lactating mothers are excluded from this study as it is unclear whether the photosensitizer sodium porfimer can cross to the feeding infant
* Patients with underlying liver disease are excluded since their metabolism of porphyrin based photosensitizers is uncertain. Evidence of liver disease will be an transaminase elevation of three times normal, a bilirubin increase of twice normal, or an alkaline phosphatase (liver fraction) elevation of twice normal.
* Patients who have underlying medical conditions that are felt to limit their survival to less than one year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2002-12; Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
The primary assessment for our first specific aim will be to determine the effect of photodynamic therapy on biomarkers after photodynamic therapy. | 12 months

SECONDARY OUTCOMES:
The primary assessment for our second specific aim will be to assess if specific biomarkers can be correlated with the confirmed histological elimination of their Barrett's esophagus. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States